CLINICAL TRIAL: NCT05776355
Title: NKG2D CAR-NK Cell Therapy for Patients With Platinum-Resistant Recurrent Ovarian Cancer
Brief Title: NKG2D CAR-NK & Ovarian Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Cheetah Cell Therapeutics Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2022-674
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Cancer
Keywords: CAR-NK
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ovarian cancer (Experimental)
  Interventions: Biological: NKG2D CAR-NK

INTERVENTIONS:
Biological: NKG2D CAR-NK — Lymphodepleting chemotherapy followed by NKG2D CAR-NK infusion

SUMMARY:
This trial will explore the maximum tolerated dose （MTD）of NKG2D CAR-NK cells in the treatment of platinum-resistant, relapsed epithelial ovarian cancer in a dose-escalation manner, and observe the clinical safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older
2. Histologically or cytologically confirmed diagnosis of epithelial ovarian cancer
3. Documented platinum resistant epithelial ovarian cancer with at least 1 measurable lesion
4. ECOG performance status of 0-2
5. Adequate organ function defined as: ANC≥1.5×109/L, PLT≥75×109/L, TBIL≤1.5×ULN, AST≤2.5×ULN, ALT≤2.5×ULN, Cr≤1.5×ULN
6. Negative urine or serum pregnancy test within 7 days prior to treatment for women of childbearing age
7. Life expectancy ≥ 12 weeks from the time of enrollment
8. All patients must have the ability to understand and willingness to sign a written informed consent form (ICF).

Exclusion Criteria:

1. Patients with history of other active malignancy within 1 year prior to enrollment;
2. Patients with central nervous system (CNS) metastases. History of any CNS disorder such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, any autoimmune disease with CNS involvement, posterior reversible encephalopathy syndrome, or cerebral edema;
3. Patients with ongoing uncontrolled serious infection, clinically significant cardiac disease (i.e., symptomatic congestive heart failure, myocardial infarction, cardiac angioplasty or stenting, unstable angina pectoris, uncontrolled cardiac arrhythmia), poorly controlled pulmonary disease (no clinically significant pleural effusion), or psychiatric illness/social situations that would limit compliance with study requirements within 12 months prior to enrollment;
4. Patients with immunologic deficiency or autoimmune diseases;
5. Known human immunodeficiency virus (HIV) seropositivity or active hepatitis B or C infection. A history of hepatitis B or C is permitted if the viral load is undetectable by quantitative assay;
6. Patients who are breastfeeding or pregnant;
7. Patients, who in the opinion of the investigator, may not be able to comply with the monitoring requirements of the study;
8. Patients participated in another investigation treatment study 4 weeks prior to enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
DLT | 28 days
  Dose-Limiting Toxicity
MTD | 28 days
  Maximal Tolerable Dose

CONTACTS AND LOCATIONS:
Overall Officials: Zhu JianQing, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No